CLINICAL TRIAL: NCT06720168
Title: Air Polishers With Erythritol in the Treatment of Dental Black Stain of Bacterial Origin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Chirag Sheth, Tenured Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCHCEU Jovani-Ribelles-Veses
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Black Stain; Black Plaque
Keywords: dental black stain; dental prophylaxis; erythritol air polisher
MeSH Terms: interventions — Dental Prophylaxis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dental prophylaxis with ultrasonic treatment (Active Comparator): Dental Prophylaxis with ultrasonics
  Interventions: Device: Dental prophylaxis with ultrasonic treatment
- Dental prophylaxis with erythritol air polishing (Experimental): Dental prophylaxis with erythritol air polishing application
  Interventions: Device: Erythritol air polisher

INTERVENTIONS:
Device: Erythritol air polisher — Dental prophylaxis with erythritol air polisher in patients with dental black stain
  Arms: Dental prophylaxis with erythritol air polishing
Device: Dental prophylaxis with ultrasonic treatment — Dental prophylaxis with ultrasonic treatment in patients with dental black stain
  Arms: Dental prophylaxis with ultrasonic treatment

SUMMARY:
Black stains on the teeth, caused by the accumulation of chromogenic microorganisms that produce iron compounds, are more common in the pediatric population and have a negative impact on dental aesthetics and patients' self-esteem. The etiology of these stains remains unclear and is not related to oral hygiene. Currently, there is no definitive treatment that prevents the reappearance of these stains, and they can only be removed by mechanical removal, which can cause injuries to the tooth structure. This study aims to evaluate the effectiveness of erythritol powder air polishers, which have antimicrobial properties, compared to conventional prophylaxis in preventing the recurrence of stains.

A randomized clinical trial will be carried out with a follow-up of 12 months, during which patient satisfaction and duration of treatment will be assessed. The results of this study could provide valuable information to improve treatment and management strategies for dental stains in the affected population, thus contributing to the emotional well-being of patients and reducing damage to their tooth enamel.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 2 or more teeth with black stain

Exclusion Criteria:

* Sistemic diseases
* Patients with physical and/or cognitive impairment which prevents participation in a dental prophylaxis.
* Use of oral antibiotics fifteen days before the intervention
* Allergy to erythritol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Recurrence of dental black stain | 3, 6, 9 and 12 months
  Following dental prophylaxis (in each of the arms) the dentist will assess the recurrence of black stains at 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Patient satisfaction | Immediately after the intervention
  Patients will received, at the end of the procedure a questionnaire to evaluate their satisfaction with the care provided, evaluating from 0 to 5 the level of disconfort experienced during the treatment (0 no disconfort, 5 maximum disconfort).

CONTACTS AND LOCATIONS:
Overall Officials: María del Mar Jovani-Sancho, DDS, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Alfara del Patriarca, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No